CLINICAL TRIAL: NCT03412162
Title: Race-based Biological Stress, Ethnic-Racial Identity, and Educational Outcomes: New Approaches to Studying Academic Achievement Gaps
Brief Title: Biology, Identity & Opportunity Study
Acronym: BIO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Harvard University (Other)
Responsible Party: Principal Investigator, Emma Adam, Edwina S. Tarry Professor and Associate Vice President for Research, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 201800033; SP0042147 (Other: Northwestern IRB)
Record Dates: First submitted 2017-12-30; First posted 2018-01-26 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Stress, Psychological; Stress, Emotional; Stress, Physiological
Keywords: Discrimination; Cortisol; Sleep; Identity
MeSH Terms: conditions — Stress, Psychological | interventions — Ethnicity

STUDY DESIGN:
Intervention Model Description: Two conditions will be tested: an ethnic-racial identity promotion intervention, and academic skills promotion control condition.
Who Masked: Outcomes Assessor
Masking Description: Post-doctoral scholar conducting the statistical data analyses will be provided with de-identified data and will not be informed of which condition is which. Rather, they will be provided with a neutral and randomly assigned set of names identifying each condition: Condition 1 and Condition 2.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ethnic and Racial Identity Promotion (Experimental): Students will participate in 8, 1 hour and 15 minute classroom based intervention sessions at their local high school, during which a facilitator will lead them through a series of lectures, group activities, and individual homework activities designed to promote a positive ethnic and racial identity (positive feelings about ones' ethnic and racial heritage and ethnic and racial group membership).
  Interventions: Behavioral: Ethnic and Racial Identity Promotion
- Academic Skills Promotion (Active Comparator): Students in this active comparison group will participate in an 8-week, 1 hour and 15 minute classroom based intervention, during which a facilitator will lead them through a series of lectures, group activities, and individual homework activities designed to provide information regarding college and career planning, and promote college and career planning as well as study skills and strategies. This condition receives the same amount of facilitator time and attention as the Experimental condition.
  Interventions: Behavioral: Academic Skills Promotion

INTERVENTIONS:
Behavioral: Ethnic and Racial Identity Promotion — See arm description
  Arms: Ethnic and Racial Identity Promotion
Behavioral: Academic Skills Promotion — See arm description
  Other Names: Attention Control Condition
  Arms: Academic Skills Promotion

SUMMARY:
This study will implement an intervention designed to promote ethnic and racial identity development. It is hypothesized that the intervention will have positive effects on ethnic-racial identity development, stress biology (including sleep hours and quality and diurnal cortisol profiles), emotional well-being, executive functioning, and academic outcomes, particularly for minority youth.

DETAILED DESCRIPTION:
On average, students from disadvantaged racial-ethnic minority groups (such as Blacks and Hispanics) show lower academic performance and attainment on a variety of measures, including grades, test scores and graduation rates. Racial-ethnic minority students are also exposed to higher levels of stress, especially "race-based stress," including higher levels of discrimination and stereotype threat. Past research has shown that race-based stress is related to alterations in stress biology, including altered stress hormone levels and less and lower quality sleep. Altered stress hormones and shorter and lower quality sleep in turn have important implications for multiple aspects of cognitive functioning, including executive functioning, that have known impacts on emotional well-being and academic performance.

It is therefore hypothesized that disparities in race-based stress and stress biology may help to account for racial-ethnic disparities in academic performance. One (correlational, non-causal) purpose of this study, therefore, is to measure and test associations among race-based social stress (RBSS, such as perceived racial discrimination), stress biology (cortisol daily rhythms and sleep hours and quality) and academic outcomes in 300 high school students in a racially diverse, mid-sized, suburban high school.

Additional research has shown that the presence of a strong ethnic-racial identity is associated with better-regulated stress biology and higher academic attainment. A second major purpose of this study, and the primary purpose of this RCT, is to test, through a random-assignment intervention, whether promoting positive ethnic and racial identity development serves to advance ethnic and racial identity development, improve stress biology, and improve emotional well-being, cognition (executive functioning), and academic outcomes. Positive effects on these outcomes are expected for those in the experimental (ethnic and racial identity promotion) group, compared to the comparison group. Effects are expected to be particularly strong for those in the experimental condition that are from black and hispanic ethnic and racial minority groups.

The present study will assess race-based social stress (received racial discrimination and stereotype threat susceptibility), ethnic and racial identity, cortisol, sleep, cognition (executive functioning), emotional and academic adjustment, and academic outcomes in a cohort of 300 high school freshman both before and after an 8-week randomized control trial of the Identity Project Intervention (Umaña-Taylor & Douglass, 2017; Umaña-Taylor, Douglass, Updegraff & Marsiglia, 2017). Participants will be recruited in 2 or (if necessary) 3 annual waves, with baseline data collection for the study starting on December 16, 2017. Initial tests of the RCT effects will occur immediately after the intervention and in the year subsequent to the intervention. Questionnaire and administrative outcomes will continue to be measured through the senior year of high school. Additional funding will be sought to measure physical health outcomes, and to follow participants into their college and/or work years. Study plans and hypotheses for these follow-on studies will be registered separately.

ELIGIBILITY:
Inclusion Criteria:

-Three hundred students will be recruited through announcements and presentations in required, non-tracked 9th grade classes at 3 mid-sized, diverse, suburban high schools, through flyers posted around the school, and through e-mails sent and presentations made to students and parent groups.

Exclusion Criteria:

* The presence of an endocrine disorder or use of corticosteroid based medications.
* Youth who are unable to read in English will be excluded because materials will solely be available in English.
* The study will not include students who do not provide parental consent.
* The study will not include students who do not provide their own assent
* The study will not include pregnant students in this study.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2017-12-16 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Ethnic and Racial Identity (ERI) development: Total Score | Within 1 month following the 8-week intervention.
  The investigators will measure an ethnic and racial identity total score from the Ethnic Identity Scale (Douglass & Umaña-Taylor, 2015). The measure uses a Likert-type scale ranging from 1 (does not describe me at all) to 4 (describes me very well). The mean score is computed for the total score. Therefore the minimum score is 1, and maximum is 4. Negatively worded items are reverse scored, so that higher scores indicate higher levels ethnic and racial identity development.
Ethnic and Racial Identity (ERI) development: Pride/Affirmation | Within 1 month following the 8-week intervention.
  The investigators will measure the ERI Pride/Affirmation subscale in the Ethnic Identity Scale (Douglass & Umaña-Taylor, 2015). The measure uses a Likert-type scale ranging from 1 (does not describe me at all) to 4 (describes me very well). The mean score is computed for the Pride/Affirmation subscale. Therefore the minimum score is 1, and maximum is 4. Negatively worded items are reverse scored, so that higher scores indicate higher levels of ethnic and racial identity pride/affirmation.
Ethnic and Racial Identity (ERI) development: Exploration | Within 1 month following the 8-week intervention.
  The investigators will measure the ERI Exploration subscale in the Ethnic Identity Scale (Douglass & Umaña-Taylor, 2015). The measure uses a Likert-type scale ranging from 1 (does not describe me at all) to 4 (describes me very well). The mean score is computed for the Exploration subscale. Therefore the minimum score is 1, and maximum is 4. Negatively worded items are reverse scored, so that higher scores indicate higher levels of ethnic and racial identity exploration.
Ethnic and Racial Identity (ERI) development: Resolution | Within 1 month following the 8-week intervention.
  The investigators will measure the ERI Resolution subscale in the Ethnic Identity Scale (Douglass & Umaña-Taylor, 2015). The measure uses a Likert-type scale ranging from 1 (does not describe me at all) to 4 (describes me very well). The mean score is computed for the Resolution subscale. Therefore the minimum score is 1, and maximum is 4. Negatively worded items are reverse scored, so that higher scores indicate higher levels of ethnic and racial identity resolution.
Ethnic and Racial Identity (ERI) development: Centrality | Within 1 month following the 8 week intervention
  The investigators will measure the centrality with a modified version of the Centrality subscale from the Multidimensional Inventory of Black Identity (MIBI; Sellers, Rowley, Chavous, Shelton, & Smith, 1997). The subscale uses a Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree). The mean score is computed for the total score. Therefore the minimum score is 1, and maximum is 7. Negatively worded items are reverse scored, so that higher scores indicate a greater extent to which a person normatively defines her or himself with regard to race. It is a measure of whether race is a core part of an individual's self-concept.
Ethnic and Racial Identity (ERI) development: Total Score | Between 9 and 12 months following the 8-week intervention.
  The investigators will measure an ethnic and racial identity total score from the Ethnic Identity Scale (Douglass & Umaña-Taylor, 2015). The measure uses a Likert-type scale ranging from 1 (does not describe me at all) to 4 (describes me very well). The mean score is computed for the total score. Therefore the minimum score is 1, and maximum is 4. Negatively worded items are reverse scored, so that higher scores indicate higher levels ethnic and racial identity development.
Ethnic and Racial Identity (ERI) development: Pride/Affirmation | Between 9 and 12 months following the 8-week intervention.
  The investigators will measure the ERI Pride/Affirmation subscale in the Ethnic Identity Scale (Douglass & Umaña-Taylor, 2015). The measure uses a Likert-type scale ranging from 1 (does not describe me at all) to 4 (describes me very well). The mean score is computed for the Pride/Affirmation subscale. Therefore the minimum score is 1, and maximum is 4. Negatively worded items are reverse scored, so that higher scores indicate higher levels of ethnic and racial identity pride/affirmation.
Ethnic and Racial Identity (ERI) development: Exploration | Between 9 and 12 months following the 8-week intervention.
  The investigators will measure the ERI Exploration subscale in the Ethnic Identity Scale (Douglass & Umaña-Taylor, 2015). The measure uses a Likert-type scale ranging from 1 (does not describe me at all) to 4 (describes me very well). The mean score is computed for the Exploration subscale. Therefore the minimum score is 1, and maximum is 4. Negatively worded items are reverse scored, so that higher scores indicate higher levels of ethnic and racial identity exploration.
Ethnic and Racial Identity (ERI) development: Resolution | Between 9 and 12 months following the 8-week intervention.
  The investigators will measure the ERI Resolution subscale in the Ethnic Identity Scale (Douglass & Umaña-Taylor, 2015). The measure uses a Likert-type scale ranging from 1 (does not describe me at all) to 4 (describes me very well). The mean score is computed for the Resolution subscale. Therefore the minimum score is 1, and maximum is 4. Negatively worded items are reverse scored, so that higher scores indicate higher levels of ethnic and racial identity resolution.
Ethnic and Racial Identity (ERI) development: Centrality | Between 9 and 12 months following the 8-week intervention.
  The investigators will measure the centrality with a modified version of the Centrality subscale from the Multidimensional Inventory of Black Identity (MIBI; Sellers, Rowley, Chavous, Shelton, & Smith, 1997). The subscale uses a Likert-type scale ranging from 1 (strongly disagree) to 7 (strongly agree). The mean score is computed for the total score. Therefore the minimum score is 1, and maximum is 7. Negatively worded items are reverse scored, so that higher scores indicate a greater extent to which a person normatively defines her or himself with regard to race. It is a measure of whether race is a core part of an individual's self-concept.

SECONDARY OUTCOMES:
Student Emotional Well-being: Student Self-Esteem | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess student emotional wellbeing, specifically student self-esteem using the Rosenberg Self-esteem Scale (Rosenberg, 1979; Phinney et al., 1997; Umaña-Taylor & Updegraff, 2007). The scale includes 10 items on a 1 (strongly disagree) through 5 (strongly agree) Likert-type scale. Five negatively worded items are reversed scored so that higher scores indicate higher levels of self-esteem. The mean score is computed for the scale. Therefore the minimum score is 1, and maximum is 5.
Student Emotional Well-being: Symptoms of Depression total score | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess student emotional wellbeing, specifically student symptoms of depression using the Center for Epidemiological Studies Depression Scale (CES-D; Hughes et al., 2004; Radloff, 1977). The CES-D includes 20 items on a 1 (rarely or none of the time) to 4 (most of the time) Likert-type scale. The CES-D consists of four subscales (Somatic Symptoms, Negative Affect, Positive Affect, Interpersonal Problems). Negatively worded items are reverse scored for the overall score so that higher scores indicate higher levels of depressive symptoms, but are not reverse scored for the positive affect subscale. A mean of the 20 items is calculated to obtain the total depressive symptoms score, therefore the minimum score is 1, and maximum is 4.
Student Emotional Well-being: Symptoms of Depression- Somatic Symptoms | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess student emotional wellbeing, specifically student symptoms of depression (somatic symptoms) using the Center for Epidemiological Studies Depression Scale (CES-D; Hughes et al., 2004; Radloff, 1977). The CES-D includes 20 items on a 1 (rarely or none of the time) to 4 (most of the time) Likert-type scale. 7 items compose the Somatic Symptoms subscale. Negatively worded items are reverse scored for the somatic symptoms subscale score, so that higher scores indicate higher levels of somatic symptoms. A mean of the 7 somatic symptoms items is calculated to obtain the Somatic Symptoms subscale score, therefore the minimum score is 1, and maximum is 4.
Student Emotional Well-being: Symptoms of Depression- Negative Affect | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess student emotional wellbeing, specifically student symptoms of depression (negative affect) using the Center for Epidemiological Studies Depression Scale (CES-D; Hughes et al., 2004; Radloff, 1977). The CES-D includes 20 items on a 1 (rarely or none of the time) to 4 (most of the time) Likert-type scale. 7 items compose the Negative Affect subscale. Negatively worded items are reverse scored for the Negative Affect subscale, so that higher scores indicate higher levels of negative affect. A mean of the 7 negative affect symptoms items is calculated to obtain the Negative Affect subscale score, therefore the minimum score is 1, and maximum is 4.
Student Emotional Well-being: Symptoms of Depression- Positive Affect | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess student emotional wellbeing, specifically student symptoms of depression (positive affect) using the Center for Epidemiological Studies Depression Scale (CES-D; Hughes et al., 2004; Radloff, 1977). The CES-D includes 20 items on a 1 (rarely or none of the time) to 4 (most of the time) Likert-type scale. 4 items compose the Positive Affect subscale. Negatively worded items are NOT reverse scored for the Positive Affect subscale, so that higher scores indicate higher levels of positive affect. A mean of the 4 positive affect symptoms items is calculated to obtain the Positive Affect subscale score, therefore the minimum score is 1, and maximum is 4.
Student Emotional Well-being: Symptoms of Depression- Interpersonal Problems | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess student emotional wellbeing, specifically student symptoms of depression (interpersonal problems) using the Center for Epidemiological Studies Depression Scale (CES-D; Hughes et al., 2004; Radloff, 1977). The CES-D includes 20 items on a 1 (rarely or none of the time) to 4 (most of the time) Likert-type scale. 2 items compose the Interpersonal Problems subscale. Negatively worded items are reverse scored for the overall score so that higher scores indicate higher levels of interpersonal problems. A mean of the 2 interpersonal problems items is calculated to obtain the Interpersonal Problems subscale score, therefore the minimum score is 1, and maximum is 4.
Student Emotional Well-being: Adolescent internalizing and externalizing total problems | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess student emotional wellbeing, specifically adolescent internalizing and externalizing symptoms using Child Behavior Check List, Youth Self Report 11-18 (CBCL YSR; Achenbach, 1991). The YSR includes 112 problem items on a 1 (not true) to 3 (very true or often true) Likert-type scale. The total problem scale is divided into 9 syndrome subscales (i.e., withdrawn, somatic complaints, anxious/depressed, social problems, thought problems, attention problems, delinquent behavior, aggressive behavior, and self-destructive/identity problems). The items are summed for a raw score, which is converted to a T-score and corresponding percentile. A T-Score of 65 or greater represents 1.5 standard deviations (or greater) above the mean, and is indicative of clinically significant adolescent problems (both internalizing and externalizing). Higher scores indicate worse symptoms.
Student Emotional Well-being: Adolescent externalizing total problems | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess student emotional wellbeing, specifically adolescent externalizing symptoms using Child Behavior Check List, Youth Self Report 11-18 (CBCL YSR; Achenbach, 1991). The YSR includes 112 problem items on a 0 (not true) to 2 (very true or often true) Likert-type scale. The externalizing problem scale can be divided into 6 syndrome subscales (i.e., social problems, thought problems, attention problems, delinquent behavior, aggressive behavior, and self-destructive/identity problems). The externalizing problems from the 6 subscales are summed for a raw score, which is converted to a T-score and corresponding percentile. T of 65 or greater represents 1.5 standard deviations (or greater) above the mean, and indicative of clinically significant externalizing problems. Higher scores are indicative of worse symptoms.
Student Emotional Well-being: Adolescent internalizing total problems | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess student emotional wellbeing, specifically adolescent internalizing symptoms using Child Behavior Check List, Youth Self Report 11-18 (CBCL YSR; Achenbach, 1991). The YSR includes 112 problem items on a 1 (not true) to 3 (very true or often true) Likert-type scale. The internalizing problem scale can be divided into 3 syndrome subscales (i.e., withdrawn, somatic complaints, and anxious/depressed). The internalizing problems from the 3 subscales are summed for a raw score, which is converted to a T-score and corresponding percentile. T of 65 or greater represents 1.5 standard deviations (or greater) above the mean, and indicative of clinically significant internalizing problems. Higher scores are indicative of worse symptoms.
Overall academic engagement | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess academic engagement using the Academic Engagement Scale (Skinner, Kindermann, & Furrer, 2008). The scale contains 10 items on a 1 (never) to 5 (all of the time) Likert-type scale. No items need to be reverse scored. Higher values indicate more engagement with school. The mean score for the 10 items is used to calculate the overall academic engagement score, with a minimum score of 1, and a maximum of 5.
Academic engagement: behavioral engagement | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess a component of academic engagement, namely, behavioral engagement, from the Behavioral Engagement subscale of the Academic Engagement Scale (Skinner, Kindermann, & Furrer, 2008). The scale contains 10 items on a 1 (never) to 5 (all of the time) Likert-type scale, and 6 items comprise the Behavioral Engagement subscale. No items need to be reverse scored. Higher values indicate more behavioral engagement with school. The mean score for the 6 items is used to calculate the behavioral engagement score, with a minimum score of 1, and a maximum of 5.
School belonging | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess school belonging, from the School Belonging Scale (McNeely, Nonnemaker, & Blum, 2002; Smalls, 2010; Smalls & Cooper, 2012). The scale contains 5 items on a 1 (strongly disagree) to 5 (strongly agree) Likert-type scale. There are no subscales in this measure. No items need to be reverse scored. Higher values reflect greater connectedness. The mean score for the 5 items is used to calculate the school belonging score, with a minimum score of 1, and a maximum of 5.
Academic motivation | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess academic motivation, from the Academic Motivation Scale (Plunkett & Bámaca-Gómez, 2003). The scale contains 5 items on a 1 (strongly disagree) to 4 (strongly agree) Likert-type scale. There are no subscales in this measure. No items need to be reverse scored. Higher values reflect more academic motivation. The mean score for the 5 items is used to calculate the academic motivation score, with a minimum score of 1, and a maximum of 4.
Academic Efficacy | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess academic efficacy, from the Academic Efficacy Scale (Alfaro et al., 2006; Alfaro et al., 2009; Midgley et al., 2000). The scale contains 5 items on a 1 (not at all true) to 5 (very true) Likert-type scale. There are no subscales in this measure. No items need to be reverse scored. Higher values reflect more academic efficacy. The mean score for the 5 items is used to calculate the academic efficacy score, with a minimum score of 1, and a maximum of 5.
Academic achievement and attainment: Standardized achievement tests | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess achievement and attainment by collecting standardized achievement tests scores, including the STAR reading and math scores.
Academic achievement and attainment: Student grades | Assessed at the end of the academic year following completion of the 8 week intervention and control curricula.
  The investigators will assess achievement and attainment by collecting student report and administrative reports on grades and collecting end of year GPA scores.
Cognition: Self-Reported Executive functioning- Global Executive Composite | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess self-reported executive functioning using the Behavior Rating Inventory of executive function Self-Report Version (Guy, Gioia, & Isquith, 2004). The BRIEF contains 80 items on a 1 (never a problem) to 3 (often a problem) Likert-type scale. The overall score for all 80 items creates the Global Executive Composite to assess an adolescent's view of his or her cognitive, emotional, and behavioral functions. The 80 items are summed for a raw score, which is converted to a T-score and corresponding percentile. T of 65 or greater represents 1.5 standard deviations (or greater) above the mean, and indicative of clinically significant deficits in executive functioning. Higher scores are indicative of worse executive functioning.
Cognition: Self-Reported Executive functioning- Behavioral Regulation Index | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess self-reported executive functioning using the Behavior Rating Inventory of executive function Self-Report Version (Guy, Gioia, & Isquith, 2004). The BRIEF contains 80 items on a 1 (never a problem) to 3 (often a problem) Likert-type scale. The Behavioral Regulation Index is comprised of 3 scales (i.e., inhibit, shift, emotional control). The items from these 3 scales are summed for a raw score, which is converted to a T-score and corresponding percentile. T of 65 or greater represents 1.5 standard deviations (or greater) above the mean, and indicative of clinically significant deficits in executive functioning, specially related to behavioral regulation. Higher scores are indicative of worse executive functioning.
Cognition: Self-Reported Executive functioning- Metacognition Index | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess self-reported executive functioning using the Behavior Rating Inventory of executive function Self-Report Version (Guy, Gioia, & Isquith, 2004). The BRIEF contains 80 items on a 1 (never a problem) to 3 (often a problem) Likert-type scale. The Metacognition Index is comprised of 5 scales (i.e., initiate, working memory, plan/organize, organization of materials, and monitor). The items from these 5 scales are summed for a raw score, which is converted to a T-score and corresponding percentile. T of 65 or greater represents 1.5 standard deviations (or greater) above the mean, and indicative of clinically significant deficits in executive functioning, specially related to metacognition. Higher scores are indicative of worse executive functioning, namely metacognition.
Cognition: Self-Reported Executive functioning- Inhibit scale | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess self-reported executive functioning (inhibition) using the Behavior Rating Inventory of executive function Self-Report Version (Guy, Gioia, & Isquith, 2004). The BRIEF contains 80 items on a 1 (never a problem) to 3 (often a problem) Likert-type scale. The Inhibit Scale is one of three scales that make up the Behavioral Regulation Index. The items from this scale are summed for a raw score, which are converted to a T-score and corresponding percentile. T of 65 or greater represents 1.5 standard deviations (or greater) above the mean, and indicative of clinically significant deficits in executive functioning, specially related to inhibition. Higher scores are indicative of worse executive functioning, namely poorer ability to control impulses (inhibitory control) and to stop engaging in a behavior.
Cognition: Self-Reported Executive functioning- Shift scale | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess self-reported executive functioning (Shifting) using the Behavior Rating Inventory of executive function Self-Report Version (Guy, Gioia, & Isquith, 2004). The BRIEF contains 80 items on a 1 (never a problem) to 3 (often a problem) Likert-type scale. The Shift Scale is one of three scales that make up the Behavioral Regulation Index. The items from this scale are summed for a raw score, which are converted to a T-score and corresponding percentile. T of 65 or greater represents 1.5 standard deviations (or greater) above the mean, and indicative of clinically significant deficits in executive functioning, specially related to shifting. Higher scores are indicative of worse executive functioning, namely poorer ability to move freely from one activity or situation to another; to tolerate change; to switch or alternate attention.
Cognition: Self-Reported Executive functioning- Emotional Control scale | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess self-reported executive functioning (Emotional Control) using the Behavior Rating Inventory of executive function Self-Report Version (Guy, Gioia, & Isquith, 2004). The BRIEF contains 80 items on a 1 (never a problem) to 3 (often a problem) Likert-type scale. The Emotional Control Scale is one of three scales that make up the Behavioral Regulation Index. The items from this scale are summed for a raw score, which are converted to a T-score and corresponding percentile. T of 65 or greater represents 1.5 standard deviations (or greater) above the mean, and indicative of clinically significant deficits in executive functioning, specially related to emotional control. Higher scores are indicative of worse executive functioning, namely poorer ability to regulate emotional responses appropriately.
Cognition: Self-Reported Executive functioning- Initiate scale | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess self-reported executive functioning (Initiation) using the Behavior Rating Inventory of executive function Self-Report Version (Guy, Gioia, & Isquith, 2004). The BRIEF contains 80 items on a 1 (never a problem) to 3 (often a problem) Likert-type scale. The Initiate Scale is one of five scales that make up the Metacognition Index. The items from this scale are summed for a raw score, which are converted to a T-score and corresponding percentile. T of 65 or greater represents 1.5 standard deviations (or greater) above the mean, and indicative of clinically significant deficits in executive functioning, specially related to initiation. Higher scores are indicative of worse executive functioning, namely poorer ability to begin an activity and to independently generate ideas or problem-solving strategies.
Cognition: Self-Reported Executive functioning- Working Memory scale | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess self-reported executive functioning (Working Memory) using the Behavior Rating Inventory of executive function Self-Report Version (Guy, Gioia, & Isquith, 2004). The BRIEF contains 80 items on a 1 (never a problem) to 3 (often a problem) Likert-type scale. The Working Memory Scale is one of five scales that make up the Metacognition Index. The items from this scale are summed for a raw score, which are converted to a T-score and corresponding percentile. T of 65 or greater represents 1.5 standard deviations (or greater) above the mean, and indicative of clinically significant deficits in executive functioning, specially related to working memory. Higher scores are indicative of worse executive functioning, namely poorer ability to hold information when completing a task, when encoding information, or when generating goals/plans in a sequential manner.
Cognition: Self-Reported Executive functioning- Plan/Organize scale | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess self-reported executive functioning (Planning/Organization) using the Behavior Rating Inventory of executive function Self-Report Version (Guy, Gioia, & Isquith, 2004). The BRIEF contains 80 items on a 1 (never a problem) to 3 (often a problem) Likert-type scale. The Plan/Organize Scale is one of five scales that make up the Metacognition Index. The items from this scale are summed for a raw score, which are converted to a T-score and corresponding percentile. T of 65 or greater represents 1.5 standard deviations (or greater) above the mean, and indicative of clinically significant deficits in executive functioning, specially related to planning/organization. Higher scores are indicative of worse executive functioning, namely poorer ability to anticipate future events; to set goals; to develop steps; to grasp main ideas; to organize and understand the main points in written or verbal presentations.
Cognition: Self-Reported Executive functioning- Organization of Materials scale | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess self-reported executive functioning (Organization of Materials) using the Behavior Rating Inventory of executive function Self-Report Version (Guy, Gioia, & Isquith, 2004). The BRIEF contains 80 items on a 1 (never a problem) to 3 (often a problem) Likert-type scale. The Organization of Materials Scale is one of five scales that make up the Metacognition Index. The items from this scale are summed for a raw score, which are converted to a T-score and corresponding percentile. T of 65 or greater represents 1.5 standard deviations (or greater) above the mean, and indicative of clinically significant deficits in executive functioning, specially related to organization of materials. Higher scores are indicative of worse executive functioning, namely poorer ability to put order in work, play and storage spaces (e.g., desks, lockers, backpacks, and bedrooms).
Cognition: Self-Reported Executive functioning- Monitor scale | Measured within 1 year of completing the 8 week intervention and control curricula.
  The investigators will assess self-reported executive functioning (Self-Monitoring) using the Behavior Rating Inventory of executive function Self-Report Version (Guy, Gioia, & Isquith, 2004). The BRIEF contains 80 items on a 1 (never a problem) to 3 (often a problem) Likert-type scale. The Monitor Scale is one of five scales that make up the Metacognition Index. The items from this scale are summed for a raw score, which are converted to a T-score and corresponding percentile. T of 65 or greater represents 1.5 standard deviations (or greater) above the mean, and indicative of clinically significant deficits in executive functioning, specially related to self-monitoring. Higher scores are indicative of worse executive functioning, namely poorer ability to check work and to assess one's own performance; ability to keep track of the effect of one's own behavior on other people.
Cognition: Executive functioning- Cognitive Flexibility and Set Switching TMT-B | Measured within 1 year of completing the 8 week intervention and control curricula.
  A brief paper and pencil measure of executive functioning, the Trail Making Test Part A (TMT-A) and B (TMT-B), will be administered (Tombaugh, 2004). TMT-B provides a measure of cognitive flexibility and set switching. The total raw score time for TMT-B is used in combination with demographic information (e.g., age, gender, education, race/ethnicity), to look up corresponding T-Scores in Heaton norms. The normal bell curve is used to evaluate T-scores (e.g., T-scores between 43 and 57 falling in the average range), with lower scores indicative of poorer executive functioning.
Cognition: Executive functioning- TMT-B total error count | Measured within 1 year of completing the 8 week intervention and control curricula.
  A brief paper and pencil measure of executive functioning, the Trail Making Test Part A (TMT-A) and B (TMT-B), will be administered (Tombaugh, 2004). TMT-B provides a measure of cognitive flexibility and set switching. The total number of errors (i.e., set-shifting and sequencing errors) for TMT-B are summed, with higher scores indicative of poorer executive functioning. The range is dependent on the number of errors made.
Cognition: Executive functioning- TMT-B set-shifting error count | Measured within 1 year of completing the 8 week intervention and control curricula.
  A brief paper and pencil measure of executive functioning, the Trail Making Test Part A (TMT-A) and B (TMT-B), will be administered (Tombaugh, 2004). TMT-B provides a measure of cognitive flexibility and set switching. The total number of set-shifting errors (i.e., not correcting shifting between letters and numbers) for TMT-B are summed, with higher scores indicative of poorer executive functioning. The range is dependent on the number of errors made.
Cognition: Executive functioning- TMT-B sequencing error count | Measured within 1 year of completing the 8 week intervention and control curricula.
  A brief paper and pencil measure of executive functioning, the Trail Making Test Part A (TMT-A) and B (TMT-B), will be administered (Tombaugh, 2004). TMT-B provides a measure of cognitive flexibility and set switching. The total number of sequencing errors for TMT-B are summed, with higher scores indicative of poorer executive functioning. The range is dependent on the number of errors made.
Cognition: Executive functioning- Cognitive Flexibility and Set Switching without basic processing speed | Measured within 1 year of completing the 8 week intervention and control curricula.
  A brief paper and pencil measure of executive functioning, the Trail Making Test Part A (TMT-A) and B (TMT-B), will be administered (Tombaugh, 2004). TMT-B provides a measure of cognitive flexibility and set switching. The total raw score time for TMT-A is subtracted from TMT-B to obtain a difference score, to remove the effects of pure processing speed from the TMT-B executive functioning scores. Higher scores are indicative of more time to complete the TMT-B task (while removing baseline processing speed), and suggestive of worse executive functioning. There are no recommended cut-offs, and this score is rather a comparative score.
Cognition: Executive functioning- Basic processing speed | Measured within 1 year of completing the 8 week intervention and control curricula.
  A brief paper and pencil measure of executive functioning, the Trail Making Test Part A (TMT-A) and B (TMT-B), will be administered (Tombaugh, 2004). TMT-A provides a measure of speed of processing. The total raw score time for TMT-A is used in combination with demographic information (e.g., age, gender, education, race/ethnicity), to look up corresponding T-Scores in Heaton norms. The normal bell curve is used to evaluate T-scores (e.g., T-scores between 43 and 57 falling in the average range), with lower scores indicative of poorer executive functioning, namely related to processing speed.
Cognition: Executive functioning, NIH Toolbox Dimensional Change Card Sort Test | Measured within 1 year of completing the 8 week intervention and control curricula.
  The NIH Toolbox Dimensional Change Card Sort Test (Gershon et al., 2013; Zelazo, & Bauer, 2013) measures set shifting, or the capacity for switching among multiple aspects of a strategy or task. Scoring is based on a combination of accuracy and reaction time. A 2-vector scoring method is employed that uses accuracy and reaction time, where each of these "vectors" ranges in value between 0 and 5, and the computed score, combining each vector score, ranges in value from 0-10. For any given individual, accuracy is considered first. If accuracy levels for the participant are less than or equal to 80%, the final "total" computed score is equal to the accuracy score. If accuracy levels for the participant reach more than 80%, the reaction time score and accuracy score are combined.
Cognition: Attention, NIH Toolbox Flanker Inhibitory Control and Attention Test. | Measured within 1 year of completing the 8 week intervention and control curricula.
  The NIH Toolbox Flanker Inhibitory Control and Attention Test (Gershon et al., 2013; Zelazo, & Bauer, 2013) measures the allocation of one's limited capacities to deal with an abundance of environmental stimulation. Scoring is based on a combination of accuracy and reaction time and is identical for both the Flanker and DCCS measures (described below). A 2-vector scoring method is employed that uses accuracy and reaction time, where each of these "vectors" ranges in value between 0 and 5, and the computed score, combining each vector score, ranges in value from 0-10. For any given individual, accuracy is considered first. If accuracy levels for the participant are less than or equal to 80%, the final "total" computed score is equal to the accuracy score. If accuracy levels for the participant reach more than 80%, the reaction time score and accuracy score are combined.
Cognition: Episodic Memory, NIH Toolbox Picture Sequence Memory Test | Measured within 1 year of completing the 8 week intervention and control curricula.
  The NIH Toolbox Picture Sequence Memory Test (Gershon et al., 2013; Zelazo, & Bauer, 2013) measures the acquisition, storage and retrieval of new information. It involves conscious recollection of information learned within a context. The PSMT is scored using IRT methodology. The number of adjacent pairs placed correctly for each of trials 1 and 2 is converted to a theta score, which provides a representation of the given participant's estimated ability in this episodic memory task. All normative standard scores are provided. Scores are converted to age-corrected Standard Scores and fully-corrected (including gender and educational level) T-Scores. The present study will use fully-corrected T-scores, which are evaluated on the normal bell curve.
Cognition: Processing Speed, NIH Toolbox Pattern Comparison Processing Speed Test | Measured within 1 year of completing the 8 week intervention and control curricula.
  The NIH Toolbox Pattern Comparison Processing Speed Test (Gershon et al., 2013; Zelazo, & Bauer, 2013) measures the amount of time it takes to mentally process a set amount of information, or the amount of information that can be processed within a certain unit of time. It is a measure that reflects mental efficiency. The participant's raw score is the number of items answered correctly in 85 seconds of response time, with a range of 0-130. This score is then converted to the NIH Toolbox normative standard scores. Scores are converted to age-corrected Standard Scores and fully-corrected (including gender and educational level) T-Scores. The present study will use fully-corrected T-scores, which are evaluated on the normal bell curve.
Cognition: Working Memory, NIH Toolbox List Sorting Working Memory Test | Measured within 1 year of completing the 8 week intervention and control curricula.
  The NIH Toolbox List Sorting Working Memory Test (Gershon et al., 2013; Zelazo, & Bauer, 2013) measures the capacity of an individual to hold information in a short-term buffer and manipulate the information. List Sorting is scored by summing the total number of items correctly recalled and sequenced on 1-List and 2-List, which can range from 0-26. This score is then converted to the nationally normed standard scores. Scores are converted to age-corrected Standard Scores and fully-corrected (including gender and educational level) T-Scores. The present study will use fully-corrected T-scores, which are evaluated on the normal bell curve.
Cognition: Fluid Intelligence | Measured within 1 year of completing the 8 week intervention and control curricula.
  The NIH Toolbox computes a Fluid Intelligence composite score (Gershon et al., 2013; Zelazo, & Bauer, 2013). This composite includes the Flanker, Dimensional Change Card Sort, Picture Sequence Memory, List Sorting and Pattern Comparison. The composite score is derived by averaging the standard scores of each of the measures, and then deriving standard scores based on this new distribution. An Age-Corrected Standard Score, Fully Corrected T-Score, Uncorrected Standard Score and associated Percentiles are computed. Higher scores indicate higher levels of functioning. An uncorrected or age-corrected standard score at or near 100 indicates ability that is average compared with others nationally. A Fully Corrected T-Score at or near 50 indicates ability that is average compared with others nationally and with similar demographic characteristics, and one below 40 suggests the possibility of health-related, acquired cognitive impairment.
Actigraphy Hours of Sleep | Measured within 1 year after completing the 8 week intervention and control curricula.
  An objective measure of hours of sleep will be determined by a research-grade actigraph, a device word on the wrist that provides an ongoing activity record that can be scored for intervals of sleeping and waking, and provide an objective estimate of total numbers of hours spent sleeping. The Sadeh scoring algorithm will be used, and hours of sleep will be examined on a scale of number of hours.
Actigraphy Sleep Efficiency | Measured within 1 year after completing the 8 week intervention and control curricula.
  An objective measure of sleep quality will be determined by actigraphy, a wristwatch-like device that provides an ongoing activity record that can be scored to provide estimates of sleep efficiency -- the proportion of time spent sleeping during the time between the individual attempted to fall asleep and their final morning awakening. Higher sleep efficiency is a reflection of better sleep quality, and is measured as a proportion or percent (on a scale from 0 to 100).
Actigraphy Sleep Latency | Measured within 1 year after completing the 8 week intervention and control curricula.
  An objective measure of sleep latency will be determined by actigraphy, a wristwatch-like device that provides an ongoing activity record that can be scored to provide estimates of sleep latency, which is the number of minutes it take from the time the individual goes to bed and when they fall asleep. Measured in number of minutes, with more minutes representing a longer sleep latency.
Cortisol: Diurnal Cortisol Slope | Measured within 1 year after completing the 8 week intervention and control curricula.
  Salivary cortisol samples self-collected by participants four times per day for four weekdays (Monday through Thursday) on the same week as the diary and sleep measurement, at waking, 30 minutes after waking, immediately after school, and at bedtime. The diurnal cortisol slope is rate of change (usually decline) in cortisol from waking to bedtime, measured in micrograms per deciliter per hour. A steeper rate of decline in cortisol from waking to bedtime is considered an indicator of positive cortisol functioning; the researchers expect a stronger decline in cortisol in the experimental as compared to the active comparison condition. The researchers expect this to be the strongest cortisol finding, with larger effect sizes than for the next two cortisol outcome variables.
Cortisol: Cortisol awakening response. | Measured within 1 year after completing the 8 week intervention and control curricula.
  Salivary cortisol samples self-collected by participants four times per day for four weekdays (Monday through Thursday) on the same week as the diary and sleep measurement, at waking, 30 minutes after waking, immediately after school, and at bedtime. The cortisol awakening response is the difference the 30 minutes post-awakening sample and the waking sample (30 minute sample - waking sample), averaged across days. The researchers expect to see a smaller cortisol awakening response among individuals in the experimental ERI intervention condition as compared to the control (active comparator) condition.
Cortisol: Average cortisol level. | Measured within 1 year after completing the 8 week intervention and control curricula.
  Salivary cortisol samples self-collected by participants four times per day for four weekdays (Monday through Thursday) on the same week as the diary and sleep measurement, at waking, 30 minutes after waking, immediately after school, and at bedtime. The average cortisol level is the area under the curve of the cortisol data points each day, divided by the total time awake that day, and averaged across the four days. This outcome will be standardized for ease of interpretation. The researchers do not expect to find significant intervention vs. control differences for this variable.

CONTACTS AND LOCATIONS:
Overall Officials: Emma K Adam, PhD, Principal Investigator — Northwestern University
Locations (3):
- United States (3):
  - Beacon Academy, Evanston, Illinois
  - District 202, Evanston, Illinois
  - District 219 Niles Township High Schools, Niles, Illinois

IPD SHARING:
Plan to Share IPD: No
Given the sensitive nature of the information and potential deductive disclosure, the investigators will only share IPD with researchers with whom they are directly collaborating, after said researchers have been added to their own (if different) and the current researchers' Institutional Review Board approval.

REFERENCES:
- [Background] Umana-Taylor AJ, Douglass S, Updegraff KA, Marsiglia FF. A Small-Scale Randomized Efficacy Trial of the Identity Project: Promoting Adolescents' Ethnic-Racial Identity Exploration and Resolution. Child Dev. 2018 May;89(3):862-870. doi: 10.1111/cdev.12755. Epub 2017 Mar 21. PMID 28321839
- [Background] Douglass, S. and A.J. Umaña-Taylor, A brief form of the Ethnic Identity Scale: Development and empirical validation. Identity, 2015. 15(1): p. 48-65.
- [Background] Umaña-Taylor, A.J., A. Yazedjian, and M. Bámaca-Gómez, Developing the ethnic identity scale using Eriksonian and social identity perspectives. Identity: An International Journal of Theory and Research, 2004. 4(1): p. 9-38.
- [Background] Rosenberg, M., Conceiving the self. New York: Basic Book. 1979: Inc.
- [Background] Phinney, J.S., The multigroup ethnic identity measure a new scale for use with diverse groups. Journal of adolescent research, 1992. 7: p. 156-176.
- [Background] Skinner, E.A., T.A. Kindermann, and C.J. Furrer, A motivational perspective on engagement and disaffection: Conceptualization and assessment of children's behavioral and emotional participation in academic activities in the classroom. Educational and Psychological Measurement, 2008.
- [Background] Guy, S.C., P.K. Isquith, and G.A. Gioia, BRIEF-SR: Behavior Rating Inventory of Executive Function--self-report Version: Professional Manual. 2004: Psychological Assessment Resources.
- [Background] Radloff, L.S., The CES-D Scale: A self-report depression scale for research in the general population. Applied Psychological Measurement, 1977. 1: p. 385-401.
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Storfer-Isser A, Lebourgeois MK, Harsh J, Tompsett CJ, Redline S. Psychometric properties of the Adolescent Sleep Hygiene Scale. J Sleep Res. 2013 Dec;22(6):707-16. doi: 10.1111/jsr.12059. Epub 2013 May 18. PMID 23682620
- [Background] Achenbach TM, Ruffle TM. The Child Behavior Checklist and related forms for assessing behavioral/emotional problems and competencies. Pediatr Rev. 2000 Aug;21(8):265-71. doi: 10.1542/pir.21-8-265. No abstract available. PMID 10922023
- [Background] Achenbach, T. M. (1991). Child Behavior Checklist/4-18. Burlington, VT: University of Vermont Department of Psychiatry.
- [Background] Gershon RC, Wagster MV, Hendrie HC, Fox NA, Cook KF, Nowinski CJ. NIH toolbox for assessment of neurological and behavioral function. Neurology. 2013 Mar 12;80(11 Suppl 3):S2-6. doi: 10.1212/WNL.0b013e3182872e5f. PMID 23479538
- [Background] Fox NA. Commentary on Zelazo and Bauer (editors), National Institutes of Health Toolbox Cognition Battery (CB): validation for children between 3 and 15 years. Monogr Soc Res Child Dev. 2013 Aug;78(4):150-5. doi: 10.1111/mono.12044. No abstract available. PMID 23952209
- [Background] Guy, S. C., Gioia, G. A., & Isquith, P. K. (2004). Behavior Rating Inventory of Executive Function-: Self-report Version. Psychological Assessment Resources.
- [Background] Tombaugh TN. Trail Making Test A and B: normative data stratified by age and education. Arch Clin Neuropsychol. 2004 Mar;19(2):203-14. doi: 10.1016/S0887-6177(03)00039-8. PMID 15010086
- [Background] Alfaro, E.C., A.J. Umaña-Taylor, and M.Y. Bámaca, The influence of academic support on Latino adolescents' academic motivation. Family Relations, 2006. 55(3): p. 279-291.
- [Background] Midgley, C., et al., Manual for the patterns of adaptive learning scales. Ann Arbor, 2000. 1001: p. 48109-1259.
- [Background] Plunkett, S.W. and M.Y. Bámaca-Gómez, The relationship between parenting, acculturation, and adolescent academics in Mexican-origin immigrant families in Los Angeles. Hispanic Journal of Behavioral Sciences, 2003. 25(2): p. 222-239.
- [Background] Umaña-Taylor AJ, Douglass S. Developing an Ethnic-Racial Identity Intervention from a Developmental Perspective: Process, Content, and Implementation of the Identity Project. In Handbook on Positive Development of Minority Children and Youth 2017 (pp. 437-453). Springer International Publishing.
- [Background] Sellers, R. M., Rowley, S. A., Chavous, T. M., Shelton, J. N., & Smith, M. A. (1997). Multidimensional Inventory of Black Identity: A preliminary investigation of reliability and constuct validity. Journal of personality and social psychology, 73(4), 805.
- [Background] Phinney, J.S., Cantu, C.L., Kurtz, D.A., 1997. Ethnic and American identity as predictors of self-esteem among African American, Latino, and White adolescents. Journal of Youth and adolescence 26, 165-185.
- [Background] Umana-Taylor AJ, Updegraff KA. Latino adolescents' mental health: exploring the interrelations among discrimination, ethnic identity, cultural orientation, self-esteem, and depressive symptoms. J Adolesc. 2007 Aug;30(4):549-67. doi: 10.1016/j.adolescence.2006.08.002. Epub 2006 Oct 23. PMID 17056105
- [Background] Hughes ME, Waite LJ, Hawkley LC, Cacioppo JT. A Short Scale for Measuring Loneliness in Large Surveys: Results From Two Population-Based Studies. Res Aging. 2004;26(6):655-672. doi: 10.1177/0164027504268574. PMID 18504506
- [Background] McNeely CA, Nonnemaker JM, Blum RW. Promoting school connectedness: evidence from the National Longitudinal Study of Adolescent Health. J Sch Health. 2002 Apr;72(4):138-46. doi: 10.1111/j.1746-1561.2002.tb06533.x. PMID 12029810
- [Background] Smalls C. Effects of mothers' racial socialization and relationship quality on African American youth's school engagement: a profile approach. Cultur Divers Ethnic Minor Psychol. 2010 Oct;16(4):476-84. doi: 10.1037/a0020653. PMID 21058810
- [Background] Smalls C, Cooper SM. Racial group regard, barrier socialization, and African American adolescents' engagement: patterns and processes by gender. J Adolesc. 2012 Aug;35(4):887-97. doi: 10.1016/j.adolescence.2011.12.007. Epub 2012 Jan 15. PMID 22248921
- [Background] Alfaro EC, Umana-Taylor AJ, Gonzales-Backen MA, Bamaca MY, Zeiders KH. Latino adolescents' academic success: the role of discrimination, academic motivation, and gender. J Adolesc. 2009 Aug;32(4):941-62. doi: 10.1016/j.adolescence.2008.08.007. Epub 2008 Oct 29. PMID 18973937